CLINICAL TRIAL: NCT05095974
Title: Echocardiography, Thoracic Fluid Content and Lung Ultrasound Monitoring as Predictors of Pulmonary Edema in Severe Preeclampsia
Brief Title: Predictors of Pulmonary Edema in Severe Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmeen alaa-eldeen elmasry, assisstant lecturer of anesthesia and intensive care, Assiut University
Other Study IDs: pulmonary edema
Record Dates: First submitted 2021-09-13; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Edema
MeSH Terms: conditions — Pulmonary Edema | interventions — Ultrasonography; Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A (main group): 29 Consecutive patients with a singleton pregnancy complicated by severe PE will be included in the study at hospital admission. Assessment will be done by lung ultrasound , echocardiography and thoracic bioimpedence device
  Interventions: Device: ultrasonography; Device: echocardiography; Device: thoracic electrical bioimpedence
- B (control group): 29 Consecutive healthy patients with a singleton pregnancy (control group) will be included in the study at hospital admission. Assessment will be done by lung ultrasound , echocardiography and thoracic bioimpedence device
  Interventions: Device: ultrasonography; Device: echocardiography; Device: thoracic electrical bioimpedence

INTERVENTIONS:
Device: ultrasonography — Ultrasound assessment will performed with parturient in the supine position using Mindray device (DC-N6, with a phased array transducer, model P4-2, 3-6 MHz). A C60x 5-2 MHz convex transducer will used for lung ultrasound (Mindray device (DC-N6, with a phased array transducer, model P4-2, 3-6 MHz).The Echo Comet Score (ECS) will obtained by the 28-rib interspaces technique dividing the chest wall in 12 areas on the left side (from the second to the fourth intercostal space) and 16 (from the second to the fifth intercostal space) on the right anterior and lateral hemithorax.
Device: echocardiography — MHz cardiac transducer for echocardiography with two-dimensional, M-mode, color-flow, continuous, pulsed wave and tissue Doppler imaging.
Device: thoracic electrical bioimpedence — EC ICONR monitor (Osypka Medical, Inc., La Jolla, California and Berlin) will be applied to the patients through four ECG electrodes. The electrodes will be placed over the bare skin of patients at the following sites: (1) on the left neck below the ear; (2) directly superior to the midpoint of the left clavicle; (3) along the left mid-axillary line at the level of the xiphoid process; (4) two-inches caudad from the third electrode.
  Other Names: electrical cardiometry

SUMMARY:
Pre-eclampsia is a multisystem major cardiovascular disease of pregnancy with hypertension its main clinical manifestation. Acute pulmonary edema, which signifies severe disease, is a leading cause of death in women with pre-eclampsia, and is a frequent cause for admission to an intensive care unit

DETAILED DESCRIPTION:
Outside pregnancy, transthoracic cardiac ultrasound (echocardiography) and lung ultrasound have become important diagnostic and monitoring tools in critically ill patients. Echocardiography allows a rapid and non-invasive assessment of myocardial contractility and preload, and lung ultrasound can be used to determine the amount of extravascular lung water (EVLW).

In pregnancy, there is evidence of a good correlation between non-invasive hemodynamic monitoring by echocardiography and invasive monitoring using a pulmonary artery catheter. Previous studies have shown that invasive hemodynamic monitoring could facilitate fluid management in patients with PE. However, recent studies have examined the utility of echocardiography in combination with lung ultrasound for guiding fluid therapy in patients with severe PE.

Thoracic fluid content (TFC) is one of the many variables measured by the ICON electrical cardiometry (EC) device (Osypka Medical, etc.). The ICON device is one relatively new proprietary implementation of impedance cardiography technology, which is also often called "thoracic electrical bio-impedance". Impedance cardiography is based on measuring the changes in total resistance of the thorax to electric current. The impedance (Zo) to electric current is determined by the resistance of different tissues such as bone, muscles, and fluids. The fluid compartment is considered the dynamic component that will cause short term changes in thoracic impedance. TFC is calculated as the reciprocal of the total thoracic impedance (1/ Zo) and is considered a numerical measure of total (intravascular and extravascular) thoracic fluid. Although TFC is a measure of both extra and intra-vascular thoracic fluid, the investigators hypothesized that it might provide an estimate of the increase in intrathoracic fluids such as to facilitate the risk of pulmonary edema.

ELIGIBILITY:
Inclusion criteria :

Pregnant women with one or more of the following:

* new-onset cerebral or visual disturbances
* thrombocytopenia (platelet count <100 000/mL)
* elevated liver enzymes (transaminases) to twice the normal upper limit;
* severe persistent pain in the right upper or middle upper abdomen that does not respond to medication and is not explained by another condition
* renal insufficiency (serum creatinine >97 μmol/L), or a doubling of serum creatinine concentration in the absence of other renal disease
* systolic blood pressure ≥160mmHg or diastolic blood pressure ≥110mmHg on more than one occasion at least 4 h apart while the patient is on bed rest (unless antihypertensive therapy had been initiated before this time).

Exclusion Criteria:

* Age below 18 yr
* SP during the postpartum period
* refusal to participate to the study.
* history of cardiac or respiratory disease
* patients with clinical manifestations of pulmonary edema

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: After obtaining approval from the Medical Research Ethics Committee Faculty of medicine, Assiut University, Assiut, Egypt, this study will be done in ICU in Assiut University Woman Health Hospital . Written informed consents will be obtained from all participants, after reading the patient information sheet and describing the procedure to the participants
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2021-10-30 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
detection of pulmonary edema | 4 days
  number of patients that will have pulmonary edema assessed by echo comet score by lung ultrasound (the sum of B-lines if yield more than 280 denoting extravascular fluid in the lung

SECONDARY OUTCOMES:
Echocardiography | 4 days
  the increase in left ventricular end-diastolic pressures measured by (E/E' ratio, E/A ratio) and left ventricular systolic function estimated by eyeball ejection fraction
Thoracic fluid content | 4 days
  the increase in thoracic fluid content measured by thoracic electrical bio-impedance device